CLINICAL TRIAL: NCT05779657
Title: Efficacy of Combined Ketamine and Midazolam for Treatment of Generalized Convulsive Status Epilepticus in Children .
Brief Title: Combined Ketamine and Midazolam for Generalized Convulsive Status Epilepticus
Acronym: Ket-Mid
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Abdelsamee Ahmed, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Soh-Med-23-03-12MS
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Generalized Convulsive Status Epilepticus
Keywords: Status epilepticus; Ketamine; Drug combination; Children; Pediatric
MeSH Terms: conditions — Status Epilepticus | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Two groups of children with continuing seizures after stabilization phase (5 minutes)
  Study group (Ket-Mid): will receive intravenous ketamine 2 mg/kg (max 60 mg) over 2 minutes.
  Control group (Pla-Mid): will receive intravenous isotonic saline (as a placebo) in the same way.
  At the same time, both groups will receive intravenous midazolam 0.2 mg/kg (maximum 10 mg) over 2 minutes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolled children will be equally randomized into study and control group using computer generated numbers, which will be sealed into sequentially numbered opaque envelopes by a person not belonging to the research team. For each enrolled participant, the envelope in order will be opened, and the assigned study drug will be used. A pharmacist will fill the active and placebo preparations in similar containers with sealed code for identification. Participants' families, treating clinicians, and investigators will be unaware of group assignment and drug/placebo therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Ket-Mid) (Experimental): Children receiving ketamine + midazolam
  Interventions: Drug: Ketamine; Drug: Midazolam
- Control group (Pla-Mid) (Placebo Comparator): Children receiving placebo + midazolam
  Interventions: Drug: Midazolam; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Intravenous ketamine 2 mg/kg (max 60 mg) over 2 minutes (diluted with isotonic saline to 5 mg/ml concentration)
  Other Names: Ketalar
  Arms: Study group (Ket-Mid)
Drug: Midazolam — Intravenous midazolam 0.2 mg/kg (maximum 10 mg) over 2 minutes
Drug: Placebo — Intravenous isotonic saline 0.4 ml/kg (max 12 ml) over 5 minutes
  Arms: Control group (Pla-Mid)

SUMMARY:
Generalized convulsive status epilepticus (GCSE) is a common neurological emergency in children. Benzodiazepines are the recommended first line antiseizure medication (ASMs), but they fail to control seizures in a third of cases. Combination of benzodiazepines with another ASM that has a different mechanism of action may be a promising option for faster control of GCSE. In this study, the investigators aim to evaluate the efficacy and safety of ketamine plus midazolam versus midazolam alone as first-line therapy of pediatric GCSE.

DETAILED DESCRIPTION:
Generalized convulsive status epilepticus (GCSE) is a common neurological emergency in children, which is associated with significant morbidity and mortality. This condition is defined as > 5 minutes of continuous or recurrent generalized tonic-clonic seizure activity without regaining consciousness. GCSE requires immediate evaluation and management in order to control ongoing seizures.

According to most guidelines, benzodiazepines are the recommended first line antiseizure medication (ASMs). Second-line ASMs for benzodiazepines-refractory GCSE include multiple options, such as fosphenytoin/phenytoin, valproic acid, or levetiracetam. Last, refractory GCSE requires treatment with third-line ASMs, such as another second-line ASMs or infusion with thiopental, midazolam, pentobarbital, propofol, or ketamine.

However, about 35% of cases with GCSE are not controlled by benzodiazepines, and up to 40% of benzodiazepines-refractory GCSE don't respond to second-line ASMs. As GCSE persists for a longer time, it becomes more difficult to control with worse prognosis. Indeed, the effectiveness of benzodiazepines to control seizures decreases by 50% when given after 10-15 minutes of continuous seizures. Therefore, new ASMs or combinations are required for earlier control of seizures, which will contribute to better outcome. Combination of benzodiazepines with another ASM that has a different mechanism of action may be a promising option for faster control of GCSE. One of the potential drugs for such combination is ketamine.

Several adult and pediatric studies have shown effectiveness of ketamine in refractory and super-refractory GCSE. Unlike benzodiazepines that act through inhibitory Gamma-aminobutyric acid (GABA), ketamine is a non-competitive antagonist for N- methyl- d- aspartate (NMDA) receptors, which mediates excitatory glutamate action. Continuous seizure activity is associated with internalization of GABA receptors and upregulation of NMDA receptors.

A number of animal studies have demonstrated synergistic action of combined ketamine and benzodiazepines for status epilepticus. While combined ketamine and benzodiazepines have been used in pediatric sedation/analgesia, there are limited studies on such combination for children with GCSE.

In this study, the investigators aim to evaluate the efficacy and safety of ketamine plus midazolam versus midazolam alone as first-line therapy of pediatric GCSE.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 month to 16 years.
* Generalized convulsive status epilepticus, defined as > 5 minutes of clinically observed continuous or recurrent generalized, tonic-clonic seizure activity without regaining of consciousness.

Exclusion Criteria:

* Failure to obtain informed consent.
* Previous treatment with any antiseizure medication for the presenting seizure episode.
* Hypertension
* Alcohol intake
* Conditions associated with increased intracranial pressure (e.g., central nervous system mass lesions, hydrocephalus)
* Glaucoma
* Known allergy or contraindications to any of the study drugs.
* End-stage kidney disease.
* End stage liver disease
* Arrhythmia, severe heart disease, or pulmonary hypertension.
* Hyperthyroidism
* Pheochromocytoma
* Hypoglycemia or hyperglycemia.
* Inborn errors of metabolism.
* Known or suspected psychiatric disorder.
* Failure to obtain intravenous access in the first 5 minutes of stabilization phase.
* Cessation of seizures during the stabilization phase (0 - 5 minutes).
* Traumatic brain injury.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Cessation of seizures at 5 minutes | 5 minutes
  Cessation of clinical seizures at 5 minutes study timepoint

SECONDARY OUTCOMES:
Need for repeating midazolam | 15 minutes
  Need for repeating midazolam during the first therapy phase
Cessation of seizures at 15 minutes | 15 minutes
  Cessation of clinical seizures at 15 minutes study timepoint
Cessation of seizures at 35 minutes | 35 minutes
  Cessation of clinical seizures at 35 minutes study timepoint
Cessation of seizures at 55 minutes | 55 minutes
  Cessation of clinical seizures at 55 minutes study timepoint
Seizure recurrence | 24 hours
  Recurrence of clinical seizures after initial cessation in the first 24 hours
Hypotension | 24 hours
  Occurrence of hypotension
Hypertension | 24 hours
  Occurrence of hypertension
Intubation | 24 hours
  Need for endotracheal intubation
Arrhythmia | 24 hours
  Occurrence of Arrhythmia
Emergence phenomenon | 24 hours
  Occurrence of emergence phenomenon, as one or more of the following: hallucination, delirium, vivid dreams, blurred/double vision, nausea/vomiting, hypersalivation.
Skin rash | 24 hours
  Occurrence of skin rash
Mortality | 24 hours
  Occurrence of death

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim A Sadek, MD, PhD, Study Chair — Faculty of Medicine, Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual patients' data will be available upon reasonable request after publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication and for 3 years
Access Criteria: Contact the principal investigator

REFERENCES:
- [Background] Trinka E, Cock H, Hesdorffer D, Rossetti AO, Scheffer IE, Shinnar S, Shorvon S, Lowenstein DH. A definition and classification of status epilepticus--Report of the ILAE Task Force on Classification of Status Epilepticus. Epilepsia. 2015 Oct;56(10):1515-23. doi: 10.1111/epi.13121. Epub 2015 Sep 4. PMID 26336950
- [Background] Singh A, Stredny CM, Loddenkemper T. Pharmacotherapy for Pediatric Convulsive Status Epilepticus. CNS Drugs. 2020 Jan;34(1):47-63. doi: 10.1007/s40263-019-00690-8. PMID 31879852
- [Background] Glauser T, Shinnar S, Gloss D, Alldredge B, Arya R, Bainbridge J, Bare M, Bleck T, Dodson WE, Garrity L, Jagoda A, Lowenstein D, Pellock J, Riviello J, Sloan E, Treiman DM. Evidence-Based Guideline: Treatment of Convulsive Status Epilepticus in Children and Adults: Report of the Guideline Committee of the American Epilepsy Society. Epilepsy Curr. 2016 Jan-Feb;16(1):48-61. doi: 10.5698/1535-7597-16.1.48. PMID 26900382
- [Background] Naylor DE. Treating acute seizures with benzodiazepines: does seizure duration matter? Epileptic Disord. 2014 Oct;16 Spec No 1:S69-83. doi: 10.1684/epd.2014.0691. PMID 25323468
- [Background] Rosati A, L'Erario M, Ilvento L, Cecchi C, Pisano T, Mirabile L, Guerrini R. Efficacy and safety of ketamine in refractory status epilepticus in children. Neurology. 2012 Dec 11;79(24):2355-8. doi: 10.1212/WNL.0b013e318278b685. Epub 2012 Nov 28. PMID 23197747
- [Background] Gaspard N, Foreman B, Judd LM, Brenton JN, Nathan BR, McCoy BM, Al-Otaibi A, Kilbride R, Fernandez IS, Mendoza L, Samuel S, Zakaria A, Kalamangalam GP, Legros B, Szaflarski JP, Loddenkemper T, Hahn CD, Goodkin HP, Claassen J, Hirsch LJ, Laroche SM. Intravenous ketamine for the treatment of refractory status epilepticus: a retrospective multicenter study. Epilepsia. 2013 Aug;54(8):1498-503. doi: 10.1111/epi.12247. Epub 2013 Jun 12. PMID 23758557
- [Background] Niquet J, Baldwin R, Norman K, Suchomelova L, Lumley L, Wasterlain CG. Midazolam-ketamine dual therapy stops cholinergic status epilepticus and reduces Morris water maze deficits. Epilepsia. 2016 Sep;57(9):1406-15. doi: 10.1111/epi.13480. Epub 2016 Aug 8. PMID 27500978
- [Background] Martin BS, Kapur J. A combination of ketamine and diazepam synergistically controls refractory status epilepticus induced by cholinergic stimulation. Epilepsia. 2008 Feb;49(2):248-55. doi: 10.1111/j.1528-1167.2007.01384.x. Epub 2007 Oct 15. PMID 17941842
- [Background] Buratti S, Giacheri E, Palmieri A, Tibaldi J, Brisca G, Riva A, Striano P, Mancardi MM, Nobili L, Moscatelli A. Ketamine as advanced second-line treatment in benzodiazepine-refractory convulsive status epilepticus in children. Epilepsia. 2023 Apr;64(4):797-810. doi: 10.1111/epi.17550. Epub 2023 Mar 2. PMID 36792542
- [Background] Sidharth, Sharma S, Jain P, Mathur SB, Malhotra RK, Kumar V. Status Epilepticus in Pediatric patients Severity Score (STEPSS): A clinical score to predict the outcome of status epilepticus in children- a prospective cohort study. Seizure. 2019 Oct;71:328-332. doi: 10.1016/j.seizure.2019.09.005. Epub 2019 Sep 11. PMID 31536850